CLINICAL TRIAL: NCT05905146
Title: Impact of a Personalized Medication Plan on Duration of Treatment With Potent Opioids in Acute Non-cancer Musculoskeletal Pain. Multicenter, Randomized, Controlled Study
Brief Title: Impact of a Personalized Medication Plan on Duration of Treatment With Potent Opioids in Acute Non-cancer Musculoskeletal Pain.
Acronym: PPPCARE II
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2020/0426/HP
Record Dates: First submitted 2023-05-23; First posted 2023-06-15 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Acute Pathology of the Locomotor System

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- interventional group (Experimental): benefiting from a multi-professional intervention around the strong opioid treatment with the aim of setting up a personalized pharmaceutical plan
  Interventions: Other: personalized pharmaceutical plan
- control group (No Intervention): routine management, including medication reconciliation at entry and exit and pharmaceutical analysis of prescriptions

INTERVENTIONS:
Other: personalized pharmaceutical plan — multi-professional intervention around strong opioid treatment with targeted pharmaceutical interview
  Arms: interventional group

SUMMARY:
The aim of this study is to evaluate whether patients who benefit from a personalized pharmaceutical plan (PPP) during their hospitalization, allowing them to be informed and sensitized, are treated for a shorter period of time with strong opioids with a reduced risk of dependence compared to a management according to the usual modalities in the rheumatology services concerned.

ELIGIBILITY:
Inclusion Criteria:

* Patient hospitalized in the rheumatology department
* Patient with acute pain in the context of a non-cancerous, non-traumatic, high-energy musculoskeletal pathology
* Patient for whom a prescription of strong opioid derivatives is initiated in rheumatology or patient for whom a prescription of strong opioid derivatives is maintained in rheumatology if the initial prescription has a maximum duration of 30 consecutive days prior to inclusion

Exclusion Criteria:

* Patient with cancer or fibromyalgia already diagnosed at inclusion
* Patient with poor French language skills
* Taking a strong opioid treatment for more than 30 consecutive days prior to inclusion
* Person judged by the prescriber or pharmacist as not autonomous for the management of strong opioid treatment
* Patient already included in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-01-18 (Actual); Primary Completion 2028-07-18 (Estimated); Study Completion 2028-07-18 (Estimated)

PRIMARY OUTCOMES:
total duration of treatment in days with strong opioids from day of inclusion | 6 months

SECONDARY OUTCOMES:
number of patients exceeding the optimal duration of treatment with strong opioids defined by the SFETD learned society (French Society for the Study and Treatment of Pain) (3 months) | 3 months
pain assessment (numerical scale) at first patient call after stopping strong opioids | 6 months
number of patients exceeding the optimal duration of treatment with strong opioids defined by the CLUD (Pain Control Committee) of Rouen University Hospital (28 days) | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Catherine CHENAILLER, Principal Investigator — University Hospital, Rouen
Locations (3):
- France (3):
  - CHU de Lille, Lille
  - CHU de Nimes, Nîmes
  - CHU de ROUEN, Rouen

IPD SHARING:
Plan to Share IPD: No